CLINICAL TRIAL: NCT05493384
Title: Telerehabilitation in Rheumatic Diseases During the Process of COVID-19 Pandemic
Brief Title: Telerehabilitation in Rheumatic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Songul Baglan Yentur, Assistant professor, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7099
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Telerehabilitation
Keywords: Telerehabilitation; Rheumatic diseases; COVID-19
MeSH Terms: conditions — Rheumatic Diseases; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): The Telerehabilitation Group will be performed exercise program including stretching, strengthening, posture and relaxation exercises by an experienced physiotherapist for 3 times a week for 8 weeks via Zoom.
  Interventions: Other: Telerehabilitation Group
- No Intervention group (No Intervention): No additional therapy will be performed to the Control Group and they were suggested to continue their usual physical activity.

INTERVENTIONS:
Other: Telerehabilitation Group — The program will include stretching, strengthening, breathing, posture, proprioceptive, relaxation exercises and segmental extremity movements. Each exercise will be performed 10 times in a session for the first 4 weeks and 15 times for the last 4 weeks. Exercises will be performed progressively on the patients.
  Arms: Telerehabilitation group

SUMMARY:
Telerehabilitation (TR) became more popular during COVID-19 pandemic due to social isolation and curfew. Exercise is one of treatments for patients with rheumatic diseases that are known to have low levels of physical activity.

DETAILED DESCRIPTION:
Telerehabilitation (TR) aims to decrease barriers such as distance, time and cost by using technology to patients and clinicians. It provides to obtain rehabilitation for patients who cannot go to a medical center due to physical, environmental or economic inadequacies. COVID-19 is a contagious respiratory disease that is caused Severe Acute Respiratory Syndrome causing Coronavirus-2 (SARS-CoV-2). It was firstly seen in December 2019 in Wuhan, China and spread rapidly all over the world. World Health Organization (WHO) was declared COVID-19 as a pandemic in March 2020. The most common symptoms are fever, cough and dyspnoea. Social isolation and staying home have been suggested to reduce the spreading rate of COVID-19 pandemic in many countries. In addition, curfew except necessity was applied in some countries and time of curfew varied by country. Patients with rheumatic diseases are at higher risk of infections because of disease activity and immunosuppression. In addition, old age and having concomitant chronic disease are among risk factors for coronavirus. Therefore, national health services recommend patients to practice self-isolation and self-quarantine. However, social isolation was concluded with more increased physical inactivity and sedentary lifestyle. Physical inactivity and disuse are proven to cause joint destruction, decreased aerobic capacity and muscle atrophy in patients with rheumatic diseases.The importance and requirement for TR were observed better during the COVID-19 pandemic. Therefore, aim of this study was to investigate the effects of TR on fatigue, depression, anxiety, sleep quality, disease activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 65
* Have diagnosed with Romatoid Arthritis, Ankylosing Spondylitis, Systemic Lupus Erthematosus or Fibromyalgia

Exclusion Criteria:

* Being pregnant
* Diagnosed with malignancy
* Had changes of medical treatment in the last 3 months
* Had dysfunction that limited physical activity such as severe neurological impairment, immobility or cooperation deficits
* Had regular exercise habit (minimally three days in a week)
* Had cardiac symphtoms according to New York Heart Association

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity scale | 2 minutes
  Fatigue is a normal response to physical exertion or stress but can also be a sign of a physical disorder. In the common sense, fatigue is a condition known to everyone from his or her own experience,irrespective of his or her age, gender, or health. Fatigue severity scale consists of nine questions; each question is scored from 1 to 7
Hospital Anxiety and Depression Scale | 2 minutes
  It consists of 14 questions that which 7 of them evaluate depression and 7 of them evaluate anxiety. Each question is scored from 0 to 3 and high scores indicate severe anxiety and depression

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index | 3 minutes
  It assesses sleep quality and disturbances over a month's time interval and consists of 19 self-rated items and five questions.It contains 7 subscales and total score is sum of these subscales. Each item is scored 0-3 and total score is changed between 0 to 21 which high scores indicate worse sleep quality.
Health Assessment Questionnaire | 2 minutes
  The questions of Health Assessment Questionnaire are about dressing and grooming, arising, eating, walking, hygiene, reach, grip and activity. The questionnaire consists of 20 questions and each question is scored from 0 to 3. Higher scores indicate worse quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home tele-rehabilitation for rheumatic patients: impact and satisfaction of care analysis — http://pubmed.ncbi.nlm.nih.gov/26945913/
- See also: Efficacy of tele-rehabilitation compared with office-based physical therapy in patients with knee osteoarthritis: A randomized clinical trial — http://pubmed.ncbi.nlm.nih.gov/26945913/